CLINICAL TRIAL: NCT02808988
Title: Effect of Periodontal Therapy and Bisphosphonates on Gingival Crevicular Fluid Levels of Nuclear Factor- κb Ligand (RANKL) and Osteoprotegerin in Postmenopausal Osteoporosis: Results of a 12-Month Study
Brief Title: Changes of GCF Levels of RANKL and Osteoprotegerin in Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Feyza Otan ÖZDEN, PhD, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: OMÜ KAEK 2012/138
Record Dates: First submitted 2016-05-27; First posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Periodontitis
Keywords: Bisphosphonate; osteoporosis; RANKL; OPG; periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Osteoporosis; Periodontitis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- group A (Active Comparator): periodontal phase 1 therapy consisted of scaling and root planning, bisphosphonate therapy (zoledronic acid), gingival crevicular fluid collection
  Interventions: Procedure: periodontal phase 1 therapy; Other: zoledronic acid
- group B (Active Comparator): periodontal phase 1 therapy consisted of scaling and root planning, no bisphosphonate therapy,gingival crevicular fluid collection
  Interventions: Procedure: periodontal phase 1 therapy
- group C (Active Comparator): no periodontal phase 1 therapy, bisphosphonate therapy (zoledronic acid), gingival crevicular fluid collection
  Interventions: Procedure: gingival crevicular fluid collection; Other: zoledronic acid
- group D (Active Comparator): no periodontal phase 1 therapy, no bisphosphonate therapy,gingival crevicular fluid collection
  Interventions: Procedure: gingival crevicular fluid collection

INTERVENTIONS:
Procedure: periodontal phase 1 therapy — periodontal phase 1 therapy consisted of scaling and root planning with ultrasonic and hand instruments under local anesthesia and gingival crevicular fluid collection by the same investigator.
  Arms: group A; group B
Procedure: gingival crevicular fluid collection — gingival crevicular fluid collection by periopapers
  Arms: group C; group D
Other: zoledronic acid — 5 mg/year zoledronic acid (i.v.)
  Arms: group A; group C

SUMMARY:
The investigators evaluated the effect of initial periodontal treatment on clinical findings and receptor activator of Nuclear Factor-kappa B ligand (RANKL) and osteoprotegerin (OPG) in gingival crevicular fluid (GCF) of patients with osteoporosis under bisphosphonate therapy within 12 months' follow-up. Clinical recordings and GCF were obtained from postmenopausal women; with chronic periodontitis and osteoporosis (Group A, n=13), with chronic periodontitis and no osteoporosis (Group B, n=12), without chronic periodontitis and osteoporosis (Group C, n=12), systemically and periodontally healthy controls (Group D, n=10) at the baseline. Recordings were repeated at the 1st, 6th and 12th months in Group A, B and C. RANKL and OPG values were measured by enzyme-linked immunosorbent assays.

DETAILED DESCRIPTION:
The study groups were selected from postmenopausal patients those referred to Department of Endocrinology, School of Medicine, Ondokuz Mayis University. Bone mineral density (BMD) measurements were performed by dual energy-X-ray absorptiometry from L1-L4 site of lumbar vertebra and/or femur (g/cm2). Osteoporosis was defined as T scores less than -2.5 at L1-L4, femur neck or total femur. Women with T scores less than -2.5 (groups A and C) were started on bisphosphonate treatment after their initial periodontal examination.

ELIGIBILITY:
Inclusion Criteria:

* Women with T scores less than -2.5 (groups A and C)
* The periodontitis patients were selected based on the radiographical evidence of bone loss, presence of four or more sites with bleeding on probing (BOP), ≥5 mm pocket depth (PD) and ≥6 mm clinical attachment loss (CAL).
* The clinically healthy control groups were selected on the basis of no radiographic bone loss or CAL and PD≤3 mm.

Exclusion Criteria:

* Any known systemic disease rather than osteoporosis
* Smoking
* Antibiotic therapy within the last 3 months
* Periodontal treatment within the last 6 months.

Ages: 50 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid levels of osteoprotegerin (OPG) and receptor activator of Nuclear Factor-kappa B ligand (RANKL) | Changes from Baseline osteoprotegerin (OPG) and receptor activator of Nuclear Factor-kappa B ligand (RANKL) at 12 months
  molecules having roles in bone resorption

CONTACTS AND LOCATIONS:
Overall Officials: Eser Sakallıoğlu, PhD,Prof.Dr., Study Director — Ondokuz Mayıs University, School of Dentistry, Department of Periodontology, Samsun, Turkey

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Anastasilakis AD, Goulis DG, Polyzos SA, Gerou S, Koukoulis G, Kita M, Avramidis A. Serum osteoprotegerin and RANKL are not specifically altered in women with postmenopausal osteoporosis treated with teriparatide or risedronate: a randomized, controlled trial. Horm Metab Res. 2008 Apr;40(4):281-5. doi: 10.1055/s-2008-1046787. Epub 2008 Feb 15. PMID 18275008
- [Result] Lane N, Armitage GC, Loomer P, Hsieh S, Majumdar S, Wang HY, Jeffcoat M, Munoz T. Bisphosphonate therapy improves the outcome of conventional periodontal treatment: results of a 12-month, randomized, placebo-controlled study. J Periodontol. 2005 Jul;76(7):1113-22. doi: 10.1902/jop.2005.76.7.1113. PMID 16018754
- [Result] Mogi M, Otogoto J, Ota N, Togari A. Differential expression of RANKL and osteoprotegerin in gingival crevicular fluid of patients with periodontitis. J Dent Res. 2004 Feb;83(2):166-9. doi: 10.1177/154405910408300216. PMID 14742657
- [Result] Bostanci N, Ilgenli T, Emingil G, Afacan B, Han B, Toz H, Atilla G, Hughes FJ, Belibasakis GN. Gingival crevicular fluid levels of RANKL and OPG in periodontal diseases: implications of their relative ratio. J Clin Periodontol. 2007 May;34(5):370-6. doi: 10.1111/j.1600-051X.2007.01061.x. Epub 2007 Mar 13. PMID 17355365
- [Result] Babur C, Ozcan G, Cebi DU, Pervane B, Ozdemir B, Yucel A, Biri AA, Babur C. Gingival crevicular fluid levels of osteoprotegerin (OPG) in premenopausal and postmenopausal women with or without chronic periodontitis. J Dent. 2012 May;40(5):364-71. doi: 10.1016/j.jdent.2012.01.013. Epub 2012 Feb 2. PMID 22326720
- [Result] Gumus P, Buduneli E, Biyikoglu B, Aksu K, Sarac F, Nile C, Lappin D, Buduneli N. Gingival crevicular fluid, serum levels of receptor activator of nuclear factor-kappaB ligand, osteoprotegerin, and interleukin-17 in patients with rheumatoid arthritis and osteoporosis and with periodontal disease. J Periodontol. 2013 Nov;84(11):1627-37. doi: 10.1902/jop.2013.120595. Epub 2013 Jan 17. PMID 23327689
- [Result] Bostanci N, Saygan B, Emingil G, Atilla G, Belibasakis GN. Effect of periodontal treatment on receptor activator of NF-kappaB ligand and osteoprotegerin levels and relative ratio in gingival crevicular fluid. J Clin Periodontol. 2011 May;38(5):428-33. doi: 10.1111/j.1600-051X.2011.01701.x. Epub 2011 Jan 24. PMID 21261673